CLINICAL TRIAL: NCT07231380
Title: Plunger Stroke Trial: A Comparison of Cyclic Manual Direct Aspiration Thrombectomy (Plunger Technique) vs. Static Manual Direct Aspiration Thrombectomy for Treatment of Acute Large Vessel Occlusion Stroke With the Raptor Aspiration Catheter
Brief Title: A Comparison of Cyclic Manual Direct Aspiration Thrombectomy (Plunger Technique) vs. Static Manual Direct Aspiration Thrombectomy for Treatment of Acute Large Vessel Occlusion Stroke
Acronym: Plunger
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Balt USA (Industry)
Responsible Party: Principal Investigator, Michael Froehler, Principle Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 251059
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke Patients; Large Vessel Occlusion
Keywords: Acute Ischemic Stroke; Large Vessel Occlusion; Mechanical Aspiration Thrombectomy; Plunger Technique; Stroke Intervention
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plunger Technique arm (Active Comparator): Participants randomized to this arm will undergo cyclic manual aspiration thrombectomy, also known as the Plunger Technique. This technique involves rhythmic, cyclic application of suction using FDA-approved devices: the Raptor Aspiration Catheter and VacLok Syringe, to remove thrombus in cases of acute ischemic stroke due to large vessel occlusion (terminal ICA or M1 segment of MCA).
  Interventions: Procedure: Plunger Technique
- Manual Static Aspiration Arm (Active Comparator): Participants randomized to this arm will undergo static manual aspiration thrombectomy, which involves continuous suction without modulation. The procedure will use FDA-approved devices: the Raptor Aspiration Catheter and VacLok Syringe, to remove thrombus in cases of acute ischemic stroke due to large vessel occlusion (terminal ICA or M1 segment of MCA).
  Interventions: Procedure: Static Manual Aspiration Thrombectomy

INTERVENTIONS:
Procedure: Plunger Technique — Rhythmic, cyclic application of suction using FDA-approved devices (Raptor Aspiration Catheter and VacLok Syringe) for clot removal in acute ischemic stroke.
  Other Names: Cyclic Manual Aspiration Thrombectomy
  Arms: Plunger Technique arm
Procedure: Static Manual Aspiration Thrombectomy — Continuous suction without modulation using FDA-approved devices (Raptor Aspiration Catheter and VacLok Syringe) for clot removal in acute ischemic stroke.
  Arms: Manual Static Aspiration Arm

SUMMARY:
This prospective, randomized controlled trial will compare two manual aspiration techniques for treating acute ischemic stroke due to large vessel occlusion: cyclic aspiration (Plunger technique) and static aspiration. Both techniques use FDA-approved devices (Raptor Aspiration Catheters and VacLok syringes) and are standard of care. Approximately 500 participants across 20 sites will be randomized to one of the two techniques. The primary endpoint is First Pass Effect (TICI 2c/3 after first attempt), with secondary endpoints including overall recanalization and 90-day functional outcomes. Results will address a critical gap in optimizing aspiration thrombectomy techniques.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, multi-center trial designed to compare two manual aspiration thrombectomy techniques for the treatment of acute ischemic stroke due to large vessel occlusion (LVO):

Cyclic Manual Aspiration (Plunger Technique): A rhythmic, cyclic application of suction, coined by Principal Investigator Dr. Michael Froehler.

Static Manual Aspiration: Continuous suction without modulation.

Both techniques will utilize FDA-approved devices, the Raptor Aspiration Catheter and VacLok Syringe which are routinely employed in clinical practice for stroke treatment. While both approaches are widely accepted, there is currently limited comparative data evaluating their relative efficacy and safety.

The study will enroll approximately 500 participants across 20 sites. Eligible patients will present with acute ischemic stroke involving the terminal internal carotid artery (ICA) or M1 segment of the middle cerebral artery (MCA). Participants will be randomized centrally in a 1:1 ratio to one of the two aspiration techniques.

Primary Endpoint:

First Pass Effect (FPE): Defined as achieving a Thrombolysis in Cerebral Infarction (TICI) score of 2c or 3 following the first attempt at clot removal.

Secondary Endpoints:

Overall recanalization rates 90-day functional outcomes (modified Rankin Scale) Successful catheter navigation to the occlusion site Procedural efficiency metrics

Both techniques are considered standard of care at Vanderbilt University Medical Center (VUMC) and other participating institutions. The study does not introduce any novel devices or untested procedures; therefore, risks to participants are minimal and comparable to routine thrombectomy procedures.

This trial addresses a critical gap in current knowledge regarding optimal manual aspiration techniques for direct aspiration thrombectomy in acute ischemic stroke. Results will provide high-quality evidence to inform best practices, potentially improving procedural efficiency and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

- Acute ischemic stroke due to occlusion of the terminal ICA or M1 segment of the MCA, Treatment can be initiated within 24 hours of symptom onset, Age 18 years or older

Exclusion Criteria:

* Evidence of acute intracranial hemorrhage prior to treatment, Failure to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
First Pass Effect (FPE) | During Procedure
  Achieving a Thrombolysis in Cerebral Infarction (TICI) score of 2c or 3 following the first attempt at clot removal.First Pass Effect (FPE):
  Thrombolysis in Cerebral Infarction (TICI) scale, ranges from 0 (no perfusion) to 3 (complete perfusion); higher scores indicate better reperfusion.

SECONDARY OUTCOMES:
Overall Recanalization Rate | During the procedure
  Achievement of successful reperfusion (TICI 2b/3) by the end of the procedure.
90-Day Functional Outcome | 90 days post procedure
  Modified Rankin Scale (mRS) score at 90 days post-procedure.Modified Rankin Scale (mRS), ranges from 0 (no symptoms) to 6 (death); higher scores indicate worse functional outcome.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jablonska M, Li J, Tiberi R, Bayraktar EA, Bilgin C, Tomasello A, Ribo M. Cyclic Aspiration in Mechanical Thrombectomy: Influencing Factors and Experimental Validation. AJNR Am J Neuroradiol. 2024 Nov 7;45(11):1708-1715. doi: 10.3174/ajnr.A8369. PMID 38844372
- [Result] Poulos DA, Keith JS, Froehler MT, Good BC. Experimental evaluation of the plunger technique: A method of cyclic manual aspiration thrombectomy for treatment of acute ischemic stroke. Interv Neuroradiol. 2024 Feb 6:15910199241230364. doi: 10.1177/15910199241230364. Online ahead of print. PMID 38321875
- [Result] Marnat G, Barreau X, Detraz L, Bourcier R, Gory B, Sgreccia A, Gariel F, Berge J, Menegon P, Kyheng M, Labreuche J, Consoli A, Blanc R, Lapergue B; ETIS Investigators. First-Line Sofia Aspiration Thrombectomy Approach within the Endovascular Treatment of Ischemic Stroke Multicentric Registry: Efficacy, Safety, and Predictive Factors of Success. AJNR Am J Neuroradiol. 2019 Jun;40(6):1006-1012. doi: 10.3174/ajnr.A6074. Epub 2019 May 23. PMID 31122921
- [Result] Kang DH, Kim BM, Heo JH, Nam HS, Kim YD, Hwang YH, Kim YW, Kim DJ, Kim JW, Baek JH, Kim YS. Effects of first pass recanalization on outcomes of contact aspiration thrombectomy. J Neurointerv Surg. 2020 May;12(5):466-470. doi: 10.1136/neurintsurg-2019-015221. Epub 2019 Sep 28. PMID 31563889
- [Result] Gross BA, Jadhav AP, Jovin TG, Jankowitz BT. Dump the pump: manual aspiration thrombectomy (MAT) with a syringe is technically effective, expeditious, and cost-efficient. J Neurointerv Surg. 2018 Apr;10(4):354-357. doi: 10.1136/neurintsurg-2017-013520. Epub 2017 Nov 10. PMID 29127194
- [Result] Arslanian RA, Marosfoi M, Caroff J, King RM, Raskett C, Puri AS, Gounis MJ, Chueh JY. Complete clot ingestion with cyclical ADAPT increases first-pass recanalization and reduces distal embolization. J Neurointerv Surg. 2019 Sep;11(9):931-936. doi: 10.1136/neurintsurg-2018-014625. Epub 2019 Feb 4. PMID 30718384
- [Result] Froehler MT. Comparison of Vacuum Pressures and Forces Generated by Different Catheters and Pumps for Aspiration Thrombectomy in Acute Ischemic Stroke. Interv Neurol. 2017 Oct;6(3-4):199-206. doi: 10.1159/000475478. Epub 2017 May 18. PMID 29118797
- [Result] Lapergue B, Blanc R, Gory B, Labreuche J, Duhamel A, Marnat G, Saleme S, Costalat V, Bracard S, Desal H, Mazighi M, Consoli A, Piotin M; ASTER Trial Investigators. Effect of Endovascular Contact Aspiration vs Stent Retriever on Revascularization in Patients With Acute Ischemic Stroke and Large Vessel Occlusion: The ASTER Randomized Clinical Trial. JAMA. 2017 Aug 1;318(5):443-452. doi: 10.1001/jama.2017.9644. PMID 28763550
- [Result] Prabhakaran S, Ruff I, Bernstein RA. Acute stroke intervention: a systematic review. JAMA. 2015 Apr 14;313(14):1451-62. doi: 10.1001/jama.2015.3058. PMID 25871671
- [Result] Campbell BCV, Donnan GA, Lees KR, Hacke W, Khatri P, Hill MD, Goyal M, Mitchell PJ, Saver JL, Diener HC, Davis SM. Endovascular stent thrombectomy: the new standard of care for large vessel ischaemic stroke. Lancet Neurol. 2015 Aug;14(8):846-854. doi: 10.1016/S1474-4422(15)00140-4. Epub 2015 Jun 25. PMID 26119323
- See also: Plunger technique — https://jnis.bmj.com/content/17/1/107

DOCUMENTS (2):
  • Study Protocol (2025-11-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT07231380/Prot_000.pdf
  • Informed Consent Form (2025-11-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT07231380/ICF_001.pdf